CLINICAL TRIAL: NCT02128152
Title: Effect of Mobility Training Using Robotic Exoskeletons on Functional Recovery in Individuals With Severe Stroke
Brief Title: Mobility Training Using Exoskeletons for Functional Recovery After Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Research Scientist, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00089523
Record Dates: First submitted 2014-02-26; First posted 2014-05-01 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Severe Stroke or Similar Neurological Muscle Weakness
Keywords: stroke; exoskeleton; Ekso; ambulation; robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ekso Training Safety and Efficacy (Experimental)
  Interventions: Device: Ekso exoskeleton

INTERVENTIONS:
Device: Ekso exoskeleton
  Other Names: Ekso by Ekso Bionics Inc.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Ekso robotic exoskeleton in persons affected by a severe stroke.

* Primary Objectives:

  * To determine if a structured high-dosage exoskeleton training program (EXTP) results in clinically significant gains in walking recovery in individuals affected by severe stroke.
  * To determine whether timing of EXTP delivery (i.e., sub-acute vs. chronic) and severity (non-ambulators vs. limited house-hold ambulators) affects the improvement in gait speed and overall function following the EXTP training protocol.
  * To determine whether maintenance or further improvement in gait speed can be achieved by an intensive follow-up program of either a traditional rehabilitation program (TRP) or extended EXTP.
* Secondary Objectives:

  * To determine the effect on functional walking endurance as assessed by the 6 minute walk test and 10 meter walk test, in high-dosage exoskeleton training program (EXTP) vs. traditional rehabilitation program (TRP) carried in an outpatient setting for post stroke individuals.
  * To determine the effect on functional balance, as assessed by the Berg Balance Scale, Functional Gait Assessment and Five times sit to stand measure as assessed by the 6 minute walk test, in high-dosage exoskeleton training program (EXTP) vs. traditional rehabilitation program (TRP) carried in an outpatient setting for post stroke individuals.
  * To determine the effect on stroke recovery, as assessed by the step counter of task specific training in high-dosage exoskeleton training program (EXTP) vs. traditional rehabilitation program (TRP) carried in an outpatient setting

DETAILED DESCRIPTION:
*Procedures During Screening Process:

This study will involve recruitment of individuals who have experienced a severe stroke as well as patients with similar neurological weakness from the inpatient setting, outpatient clinics, as well as day rehabilitation sites through The Rehabilitation Institute of Chicago and Northwestern Memorial Hospital.

Members of the research team will perform the initial screening of potential subjects. These clinicians will determine study eligibility based on the inclusion and exclusion criteria provided by Ekso Bionics in accordance with the medical recommendations of Dr. Todd Kuiken.

Potential subjects will be asked questions regarding their medical history and current level of function. If the subject meets the criteria, researchers will then provide the subject with a consent form. The researchers will discuss the objectives, study protocol, and the risks and benefits of the study with each subject. The subjects will be given time to review the form and ask any questions about the study.

Once each subject has provided informed consent, he or she will undergo a screening process to assess joint range of motion, muscular strength (via manual muscle test), and any spasticity present (via Modified Ashworth Scale). These measures will be used to determine subject qualification based on inclusion and exclusion criteria. Vital signs (including heart rate, blood pressure and oxygen saturation) will be assessed at baseline, after each session, and during sessions as needed based on subject's signs and symptoms. Oxygen saturation and heart rate will be monitored using a pulse oximeter. Blood pressure will be assessed with a manual blood pressure cuff and stethoscope.

*Procedures During Treatment:

Sessions will begin with donning the Ekso device to ensure a proper fit. A physical therapist will check the subject for proper alignment of joints with the device and check for areas of increased pressure between the device and body. If necessary, additional padding will be added to ensure safety and comfort or the device configuration will be modified. During the initial sessions, skin checks will be more frequent as padding is customized, after which they will occur at the end of each session.

After the pre-session measures, the participant will be attached to a suspension device (Guldman overhead lift) and guarded by facility clinical/Ekso Bionics staff to ensure participant safety. Each participant will undergo measurement, sizing, and donning of the Ekso device in addition to skill training. Each participant will then be instructed in proper use of the Ekso device and progressed through a series of weight shifting, balance, and walking skill sets. Participants will be scheduled for an initial screening session and up to 26 follow-up training sessions and assessments after the 9th, 18th, and 26th session. A follow-up assessment will also take place 3 months after the 26th training session. The amount of sessions provided will be dependent upon compatibility with device, ability to tolerate device use, and ability to safely ambulate using the device. A participant will continue with each phase of the study as deemed appropriate by research staff:

* Phase 1 (1-9 training sessions): Each subject will be instructed in regards to optimal postural alignment and weight shifting strategies to walk more efficiently in the device. The subject will complete balance and weight shifting tasks to improve standing balance and initiation of stepping in the device. Each subject will participate in 90 minute gait training sessions with an emphasis multi-directional weigh shifting, balance, and initial walking tasks in the device.
* Phase 2 (10-18 training sessions): Each subject will continue with gait training in the Ekso device utilizing training protocols developed to achieve progression with walking from maximum-assist, tethered walking towards a greater level of independence including non-tethered walking in the device. An assessment of gait speed, among other functional measures, will take place during the 18th session. Each subject's gait speed will determine the type of training that he or she will receive during the sessions 19-26.
* Phase 3 (19-26 training sessions): Subjects with a walking speed <.4m/sec will continue with Ekso device gait training for 4 weeks at a rate of 2 sessions per week. Subjects with a walking speed of >.4m/sec will continue with traditional physical therapy treatment for 4 weeks at a rate of 2 sessions per week. Both types of training sessions will focus on improving overall balance, walking distance, walking speed, & confidence with over ground walking.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be post stroke or have similar neurological weakness (2 weeks up to 6 months post and 6 months or more post)
* Subjects must be between 18-85 years of age
* Subjects must be able to fit into device and have joint motion to allow ambulation in device
* Subjects must be able to tolerate upright standing for 30 minutes
* Subjects must have sufficient upper extremity strength and balance to allow ambulation with device
* Subjects must have walking speed <0.4m/s, including non-ambulators
* Subjects must be able and willing to give written consent and comply with study procedures, including follow-up visits
* Mini Mental Status Exam (MMSE) score >17
* Medical clearance from physician

Exclusion Criteria:

* Subjects must not be shorter than 60 inches or taller than 74 inches
* Subjects must not weight greater than 220 lbs
* Joint contractures of the hip, knee, or ankle that might limit normal ROM during ambulation
* Medical issue that precludes full weight bearing and ambulation (e.g. orthopedic injuries, pain, severe osteoporosis, or severe spasticity)
* History of significant problems with skin breakdown or current skin breakdown that would prevent subject from wearing the device
* Cognitive and/or communicative disability (e.g. due to brain injury). Patients must be able to follow directions and demonstrate learning capability
* Pregnancy
* Untreated deep vein thrombosis (DVT)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in 6 Minute Walk Test With VO2 Analysis | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The 6MWT measures the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The minimal detectable change distance for people with sub-acute stroke is 60.98 meters15. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. This test will be administered while wearing a mask to measure oxygen consumption.
Change in 10 Meter Walk Test | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  This test will examine the patient's gait speed. Patients will be directed to walk at their preferred maximum but safe speed. Patients will be positioned 1 meter before the start line and instructed to walk the entire distance and past the end line approximately 1 meter. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundredth of a second (ex: 2.15 sec). The test will be recorded 2 times, with adequate rest in between. The average of the 2 times should be recorded.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Assessment of Motor Recovery After Stroke | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The purpose of the FMA is to evaluate and measure recovery in post-stroke hemiplegic patients. There are five domains assessed on a 3 point ordinal scale from 0-2. "0" is equal to "cannot perform", "1" is equal to "performs partially", and "2" is equal to "performs fully. The domain for lower extremity motor function will be used.
Change in Mini Mental Status Examination | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The MMSE is a brief screening tool used to provide a quantitative evaluation of cognitive impairment. MMSE briefly measures orientation to time and place, immediate recall, short-term verbal memory, calculation, language, and construct ability.
Change in Modified Falls Efficacy Scale | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The mFES is a 14 item self-report survey that assesses an individual's perception of balance and stability during indoor and outdoor activities of daily living. The mFES is a 10 point numerical rating scale with higher scores indicating higher confidence in the performance of the activity.
Change in Activities Specific Balance Confidence Scale | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The ABC is a 16-item self-report questionnaire that measures confidence in performing various ambulatory activities without falling. Items are rated on a scale ranging from 0-100, with zero representing no confidence and 100 representing complete confidence. It has good to excellent reliability and adequate construct validity, correlating with the BBS and 10mWT.
Change in Community Participation Indicators | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The CPI is an eighty-item self-report questionnaire that assesses the individual's satisfaction with their community participation.
Change in Visual Analog Scale | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The 0-10 rating scale for pain is used to gain a subjective report of the intensity of a person's pain. Zero represents "no pain" and ten represents "the most intense pain imaginable". A meaningful change would be plus or minus 3 points.
Change in The Psychosocial Impact Of Assistive Devices Scale | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The PIADS is 26 item questionnaires used to assess the impact assistive devices have on the quality of life of an individual who utilizes them. The questionnaire is composed of three subscales: competence, self-esteem, and adaptability. Each item is scored on a 7 point scale with a negative number indicating negative impact and a positive number indicating a positive impact.
Change in Patient Health Questionnaire-9 | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The PHQ-9 is a 9-item self-report screening assessment for depression. It is the depression module of the Diagnostic and Statistical Manual (4th edition). Each item is scored from 0-3; total scores may be 0-27, with higher scores representing increased severity of depression.
Change in Stroke Specific Quality of Life | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The SSQoL is a self-report questionnaire that is accepted as a reliable and valid way to assess health-related quality of life specific to stroke survivors. Subjects respond to 49 questions in 12 domains: mobility, energy, upper extremity function, work/productivity, mood, self-care, social roles, family roles, vision, language, thinking, and personality. Each item is rated on a 5-point Likert scale, with higher scores indicating better functioning. Domains scores (un-weighted average of item scores) and a summary score (un-weighted average of all 12 domain scores) are computed.
Change in Range of Motion | Session 1 (pre test, initial visit) and Session 32 (post test, 10 weeks)
  Range of motion of the joints of the upper and lower extremities will be measured using a goniometer.
Change in Manual Muscle Test | Session 1 (pre test, initial visit) and Session 10 (post test, 10 weeks)
  Manual muscle testing is a procedure for the evaluation of the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance.
Change in Modified Ashworth Test | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The Modified Ashworth Scale is a 6 point ordinal scale used to grade the amount of hypertonicity in individuals with neurological diagnoses. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner.
Change in Stops While Walking Test | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The SWWT can be used to determine the effects of attentional demands during walking by introducing a secondary task, talking, while walking. The subject walks at a pre-selected comfortable speed. Yes or no questions are asked while the subject is walking. The test is positive if the subject stops or demonstrates deviations at a result of talking while walking.
Change in Berg Balance Scale | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The BBS is a 14-item objective measure designed to assess static balance and fall risk in adult populations and is a well-accepted measure in the stroke literature. The functional activities that are assessed include sitting and standing balance during transfers, altered base of support, reaching, turning, eyes open and closed. Each item is scored from 0 to 4 points. The maximum score is 56 points. A score from 0 to 20 represents balance impairment, 21 to 40 represents acceptable balance, and 41-56 represents good balance.
Change in 5 Times Sit to Stand Test | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The 5xSST is used to measure functional lower extremity strength during the transitional movement of sit to stand. The individual is timed in moving from the start position of sitting, arms across chest, in a standard chair without armrests to fully standing five times.
Change in Timed Up And Go | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The TUG is a timed test used to assess mobility, balance, and walking in people with balance impairments. The subject must stand up from a chair (which should not be leaned up against a wall), walk a distance of 3 meters, turn around, walk back to the chair and sit down - all performed as quickly and as safely as possible.
Change in Functional Reach Test | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The Functional Reach test is used to objectively measure a person's stability by measuring the distance an individual can reach forward while standing without taking a step. This is performed three times. The results of the last two trials are averaged to determine the result of the exam.
Change in Modified Functional Reach | Session 1 (pre test, initial visit), Session 12 (week 4), Session 22 (week 7), Session 10 (post test, 10 weeks) and Session 33 (3 month follow-up visit)
  The Modified Functional Reach test is used to assess the stability of individuals who cannot stand by measuring the distance they can reach forward while sitting without rotating. This is performed in three different standard positions three times each with a 15 second rest break between each trial. The results of the last two trials in each direction are averaged to determine the result of the exam.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States